CLINICAL TRIAL: NCT07320079
Title: Evaluation of the Effectiveness of Health Literacy Education Given to Women by Teach-Back Method: Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness of Health Literacy Education Given to Women by Teach-Back Method
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Fatma Dünmez, PhD student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-708
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Health Literacy; Teach Back
Keywords: Health literacy; Teach-back; Women; Self-efficacy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental group and control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach-back (Experimental): The experimental group will receive face-to-face health literacy education using the teach-back method in six sessions, each lasting 45 minutes per week.
  The training will be provided by the researcher on a one-to-one basis. Health literacy education will be delivered using the teach-back method. After each session, participants will be asked to repeat what they have learned in their own words. The researcher will assess how well the participants have understood the topic. Any misunderstandings will be identified and corrected. During this process, participants will also have the opportunity to ask questions. Additional information will be provided if necessary until participants can accurately repeat the expected knowledge. The module will be considered complete once the participants have correctly expressed the information and understood the topic. The following week, the next module will begin, and this process will continue until all six modules are completed.
  Interventions: Other: teach-back
- Control Group (Other): The control group will receive standard care.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: teach-back — The experimental group will receive face-to-face health literacy education using the teach-back method in six sessions, each lasting 45 minutes per week.
  The training will be provided by the researcher on a one-to-one basis. Health literacy education will be delivered using the teach-back method. After each session, participants will be asked to repeat what they have learned in their own words. The researcher will assess how well the participants have understood the topic. Any misunderstandings will be identified and corrected. During this process, participants will also have the opportunity to ask questions. Additional information will be provided if necessary until participants can accurately repeat the expected knowledge. The module will be considered complete once the participants have correctly expressed the information and understood the topic. The following week, the next module will begin, and this process will continue until all six modules are completed.
  Arms: Teach-back
Other: Control Group — The control group will receive standard care
  Arms: Control Group

SUMMARY:
This study aims to enhance women's health literacy levels and to examine the effectiveness of the teach-back teaching technique in improving women's health literacy. The research was designed as a randomized controlled study. In addition, this study aims to answer the question of whether health literacy education delivered using the teach-back method is effective in improving women's health literacy levels. Within the scope of the study, participants in the experimental group will receive health literacy education using the teach-back technique, while the control group will receive standard care. Data will be collected using a questionnaire method.

DETAILED DESCRIPTION:
This study aims to enhance women's health literacy levels and to examine the effectiveness of the teach-back teaching technique in improving women's health literacy. Women aged between 18 and 65 years with a General Health Questionnaire-12 score below 4 will be included in the study. To determine the participants' socio-demographic and health characteristics, the "Personal Information Form" will be used; to assess general health, the "General Health Questionnaire-12" will be applied; to measure health literacy levels, the "Türkiye Health Literacy Scale-32 (TSOY-32)" will be utilized; and to assess self-efficacy, the "General Self-Efficacy Scale" will be employed. Additionally, the "Training Effectiveness Evaluation Form" will be used to evaluate the effectiveness of the education provided to the experimental group. The study will consist of a total of 74 participants, with 37 in the experimental group and 37 in the control group. Verbal and written consent will be obtained from participants who agree to take part in the study, and the participants will be assigned to groups accordingly. The experimental group will receive face-to-face health literacy education using the teach-back method in six sessions, each lasting 45 minutes per week. The control group will receive standard care.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 65 years
* Those with a General Health Questionnaire-12 score below 4

Exclusion Criteria:

* Illiterate women
* Male individuals
* Those with communication difficulties
* Healthcare professionals (physicians, midwives, nurses, etc.)
* Emergency patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Health literacy | Measurements will be taken at baseline, immediately after the training (week 6), and one month after the training (week 10).
  The Turkey Health Literacy Scale-32 will be used to measure health literacy levels. It is a scale consisting of 32 questions. The total score takes values between 0 and 50. 0 indicates the lowest health literacy level, and 50 indicates the highest health literacy level.
  According to the scoring system below, health literacy is defined as follows:
  a score of 0-25 indicates inadequate health literacy; a score of >25-33 indicates problematic-limited health literacy; a score of >33-42 indicates adequate health literacy; and a score of >42-50 indicates excellent health literacy.
The General Self-Efficacy Scale | Measurements will be taken at baseline, immediately after the training (week 6), and one month after the training (week 10).
  The General Self-Efficacy Scale will be used to measure the participants' self-efficacy levels. The scale is a 5-point Likert-type instrument consisting of three subdimensions and 17 items. The subdimensions are Initiation (9 items), Persistence (5 items), and Maintenance Effort-Determination (3 items). The total scale score ranges from 17 to 85, with higher total scores indicating a higher level of self-efficacy belief.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No